CLINICAL TRIAL: NCT01834001
Title: Evaluation of Local Response of Prostate Cancer to Irradiation Using Multiparametric MRI and MR-Guided Biopsies
Brief Title: Imaging Studies to Check the Local Response of Prostate Cancer to Radiation Therapy
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130119; 13-C-0119
Record Dates: First submitted 2013-04-13; First posted 2013-04-17 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-14

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Prostatic Neoplasms; Radiation; Biochemical Failure; Natural History
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Untreated prostate cancer: Patients with untreated prostate cancer
- 2/Radiotherapy treated prostate cancer: Patients with prostate cancer who have already received definitive radiotherapy and have experienced biochemical failure

SUMMARY:
Background:

- Radiation is a common treatment for prostate cancer. It helps damage tumor cells and causes them to die. Radiation can be effective, but some tumors may be harder to treat with radiation or even with surgery. This happens to a small number of men who have either radiation or surgery for prostate cancer. Most men who have these hard-to-treat tumors do not know if the tumor has recurred only in the prostate or has spread to another area. Also, men whose prostate cancer has recurred only after radiation may have different treatment options. This study will use improved imaging studies to better understand why some men do not respond as well to initial radiation treatments.

Objectives:

- To use detailed imaging studies to look at the results of local radiation therapy for prostate cancer.

Eligibility:

* Men at least 18 years of age who are scheduled to have radiation for prostate cancer.
* Men at least 18 years of age whose prostate cancer has returned after earlier treatments.

Design:

* All participants will have a medical history and physical exam. Blood and urine samples will be collected. Imaging studies will be used to evaluate the cancer at the start of the study.
* All participants will have an initial full magnetic resonance imaging (MRI) scan of the prostate. Tumor and healthy tissue samples will be collected.
* Those whose cancer has recurred after treatment will discuss possible treatment options with the study doctors.
* Participants who are scheduled to have radiation will have radiation therapy. This will be given according to the current standard of treatment.
* After radiation, participants will have regular follow-up tests and imaging studies. They will have another full MRI scan 6 months after the end of radiation treatment.

DETAILED DESCRIPTION:
Background:

Radiation therapy is a commonly used therapy for prostate cancers. The majority of men with prostate cancer will be cured by therapy; however, a subset, typically men with bulky or higher risk disease will develop PSA failure after definitive radiotherapy.

Currently, men with a rising PSA after radiotherapy may receive hormonal therapy or may undergo further evaluation for local failure.

It is not known how many men with rising PSA after radiotherapy may have a local failure and would benefit from a salvage local therapy. With the availability of a growing number of local salvage options, accurately defining the presence and characteristics of local failure is critical.

Objective:

To determine the rate of local recurrence in patients with prostate cancer treated with radiotherapy using multiparametric prostate MR guided and standard biopsies.

Eligibility:

Patients with no local therapy for prostate cancer:

Age >= 18 years.

Histologically confirmed adenocarcinoma of the prostate.

Intermediate or high risk prostate cancer (clinical stage >=T2b, Gleason score 7 or higher, or PSA >10, extracapsular extension or seminal vesicle invasion on MRI).

Patient will be treated with radiotherapy for prostate cancer.

ECOG performance status <=2.

Patients with biochemical relapse after radiotherapy for prostate cancer:

Evidence of prostate cancer recurrence (palpable abnormality after radiotherapy, radiographic evidence of local failure, biochemical relapse).

ECOG performance status <=2.

Age >= 18 years.

Histologically confirmed adenocarcinoma of the prostate.

Design:

Patients with untreated prostate cancer:

Participants will be screened with a physical examination, medical history, laboratory tests (CBC, chemistries, liver transaminases, PSA, PT/PTT), and imaging studies (as appropriate to staging).

Patients will undergo multiparametric MR imaging and MR guided prostate biopsy of all suspicious lesions (diagnostic and research).

Patients will receive radiotherapy at NIH or at an outside facility.

Patients will return for follow up at 3 month intervals for the first 2 years and then every six months for 5 years for PSA measurement.

Patients will undergo a multiparametric MR at 6 months after therapy. No biopsy is obtained unless patients meet the definition of treatment failure. This study would allow future correlation with early changes that may predict for eventual outcome.

Patients with a rising PSA that meet the criteria for biochemical failure by the Phoenix definition will undergo repeat multiparametric prostate MRI with biopsy of suspicious lesions (diagnostic and research).

Patients with recurrent prostate cancer:

Participants will be screened with a physical examination, medical history, laboratory tests (CBC, chemistries, Liver transaminases, PSA, PT/PTT), and imaging studies.

Patients will undergo multiparametric MR imaging and MR guided prostate biopsy of all suspicious lesions (diagnostic and research).

120 patients with untreated prostate cancer and 100 patients with biochemical recurrence after radiotherapy will be accrued to this study.

ELIGIBILITY:
* INCLUSION CRITERIA: men with untreated prostate cancer.

  1. Patients must have histologically or cytologically confirmed prostate cancer. The outside pathology report is acceptable for study entry. Every effort will be made to acquire the outside pathology slides to be confirmed by the Laboratory of Pathology, NCI.
  2. Intermediate or high risk prostate cancer (clinical tumor stage T2b or higher, Gleason 7 or higher, or PSA greater than 10). Previously obtained MR imaging may be used for clinical T staging (extracapsular extension, seminal vesicle invasion).
  3. No prior local therapy (prostatectomy, radiation, cryotherapy) or hormonal therapy for prostate cancer.
  4. Age >18 years.
  5. ECOG performance status <2 (Karnofsky >60%).
  6. Radiotherapy is planned as definitive therapy for prostate cancer. For patients not treated at NCI ROB patients must have a radiation oncologist who is willing to collaborate with the ROB and provide documentation of treatment.
  7. Ability of subject to understand and the willingness to sign a written informed consent document.

INCLUSION CRITERIA: for men with presumed prostate cancer relapse

1. Patients must have a history of histologically or cytologically confirmed prostate cancer. The outside pathology report is acceptable for study entry. Every effort will be made to acquire the outside pathology slides to be confirmed by the Laboratory of Pathology, NCI
2. Age greater than or equal to 18 years.
3. ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
4. Radiotherapy (external beam irradiation alone or in combination with hormonal therapy and/or brachytherapy) was delivered as definitive therapy for prostate cancer and documentation is available.
5. Evidence of prostate cancer recurrence (biochemical relapse by the Phoenix definition, enlarging palpable prostatic abnormality, imaging evidence strongly suggestive of local failure)
6. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients unable to tolerate MRI (patients with pacemakers, cerebral aneurysm clips, shrapnel injuries, or other implantable electronic devices or metal not compatible with MRI).
2. Evidence of metastases (pelvic lymph node involvement is not an exclusion criteria). For patients with recurrent prostate cancer, oligometastatic disease (3 or fewer visible metastases) is not an exclusion criterion.
3. Patients with coagulopathies who are at increased risk for bleeding or on active anticoagulation therapy (platelets less than 100,000 per mm^3 or PT/PTT greater than 1.5 times the upper normal limit (UNL). Patients are eligible if the underlying cause is correctable.
4. Subject s weight exceeding MRI or radiation treatment table tolerance.
5. Patients with active urinary tract infections.
6. Patients with renal insufficiency with a GFR less than 30, due to the fact that they will not be able to undergo gadolinium enhanced MRI.
7. Uncontrolled illness or comorbidity that in the judgment of the PI would preclude participation in the study.
8. Hepatitis B or Hepatitis C active infection.
9. HIV-positive patients are ineligible because HIV is known to increase radiation toxicity and may result in under-dosing or alterations in the treatment plan that would alter the likelihood of local recurrence. Appropriate studies will be undertaken in HIV positive patients when indicated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with untreated prostate cancer and men with presumed prostate cancer relapse
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-11-13 (Actual); Primary Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
To determine the rate of local recurrence in patients with prostate cancer treated with radiotherapy using multiparametric prostate MR -guided and standard biopsies. | completion of study
  The primary objective is to determine the rate of local recurrence in patients with intermediate and high risk prostate cancer treated with radiotherapy that develop a rising PSA.

SECONDARY OUTCOMES:
Post-treatment Multiparametric MR imaging | completion of study
  To determine if post-treatment multiparametric MR imaging correlates with treatment effect or pathologic grade on biopsy
MR images at failure | completion of study
  To compare MR images obtained at failure to whole mount prostate pathology in patients who undergo eventual salvage prostatectomy
Local failure detection | completion of study
  To determine if prostate MR and MR-guided biopsies enhance the ability to detect local failure after radiation compared to standard biopsy alone.
clinical and radiographic predictors of local recurrence | completion of study
  To determine the pre-treatment clinical and radiographic predictors of local recurrence in intermediate and high risk prostate cancer patients treated with radiotherapy
Changes in tumor tissue | completion of study
  To evaluate changes in tumor tissue from post-radiotherapy recurrence compared to pre-treatment biopsies with the goal of defining factors of radiation resistance
Biologic predictors of local recurrence | completion of study
  To define biologic predictors of local recurrence in intermediate and high risk prostate cancer patients treated with radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. @@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0119.html